CLINICAL TRIAL: NCT01520857
Title: A Controlled Randomized Trial Comparing Spinal Versus General Anesthesia for Transabdominal Preperitoneal (TAPP) Repair of Inguinal Hernia
Brief Title: Spinal Versus General Anesthesia for Transabdominal Preperitoneal (TAPP) Repair of Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Chamaidi Sarakatsianou, RN,MSc, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTH5535/12/11
Record Dates: First submitted 2012-01-19; First posted 2012-01-30 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Postoperative Pain
Keywords: Laparoscopic inguinal hernia repair; TAPP; Spinal Anesthesia; General Anesthesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinal anesthesia (Active Comparator): Transabdominal Preperitoneal repair of inguinal hernia. spinal anesthesia
  Interventions: Procedure: Transabdominal Preperitoneal repair of inguinal hernia
- General Anesthesia (Active Comparator): Transabdominal Preperitoneal repair of inguinal hernia. general anesthesia
  Interventions: Procedure: Transabdominal Preperitoneal repair of inguinal hernia

INTERVENTIONS:
Procedure: Transabdominal Preperitoneal repair of inguinal hernia — Transabdominal Preperitoneal (TAPP) repair of inguinal hernia using CO2 pneumoperitoneum under spinal anesthesia
  Arms: Spinal anesthesia
Procedure: Transabdominal Preperitoneal repair of inguinal hernia — Transabdominal Preperitoneal (TAPP) repair of inguinal hernia using CO2 pneumoperitoneum under general anesthesia
  Arms: General Anesthesia

SUMMARY:
The purpose of the study is to assess whether spinal anesthesia is superior to the standard general anesthesia or not for patients undergoing transabdominal preperitoneal inguinal hernia repair (TAPP).

DETAILED DESCRIPTION:
Anesthesia for laparoscopic procedures, including transabdominal preperitoneal inguinal hernia repair(TAPP) is synonymous with general anesthesia because of the adverse effects of the CO2 pneumoperitoneum on the awake patient, and regional anesthesia is preferred only in patients where general anesthesia is contraindicated. Α pilot study of our hospital has recently shown the feasibility to perform successfully and safely transabdominal preperitoneal inguinal hernia repair with low pressure CO2 pneumoperitoneum under spinal anesthesia.After this pilot study and based on previous experience in regional anesthesia for laparoscopic procedures, we designed a controlled randomized trial in order to compare spinal anesthesia with the standard general anesthesia for patients undergoing transabdominal preperitoneal inguinal hernia repair (TAPP).

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* BMI ≤ 35
* Age ≥ 18
* Normal coagulation profile

Exclusion Criteria:

* Non-reducible/obstructed hernias
* Previous open surgery in the lower abdomen
* Contraindication for pneumoperitoneum
* Contraindication for spinal or/and general anesthesia
* History of chronic pain or daily intake of analgesics
* Psychiatric disorders
* Inability of patients to use PCA pump

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | Every 8 hours
  The total dose of morphine was calculated as mg and administered by PCA pump

SECONDARY OUTCOMES:
Postoperative pain | Every 8 hrs
  NRS = numeric rating scale 0-10 mm (0=no pain to 10= worst imaginable pain)
Side- effects | Every 8 hrs
  To determine the occurrence of side effects such as postoperative nausea,vomiting, itching, headache, shoulder pain, urinary retention, etc
Hospital stay | Patients will be followed for the duration of hospital stay
Patient satisfaction | 2 weeks after the operation
Chronic Pain | 12 months after the operation
Quality of life | 6 months after the operation
  SF 36 questionnaire
Complications | 1 year
  seroma, hematoma, infection, recurrence of hernia, etc

CONTACTS AND LOCATIONS:
Overall Officials: Chamaidi Sarakatsianou, RN,MSc, Principal Investigator — University Hospital of Larissa; George Tzovaras, MD, Study Chair — University Hospital of Larissa; George Tzovaras, MD, Study Director — University Hospital of Larissa; Stavroula Georgopoulou, MD, Study Director — University Hospital of Larissa
Locations (1):
- University Hospital of Larissa, Larissa, Greece